CLINICAL TRIAL: NCT01100775
Title: Effects of Galantamine on Cognition
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, L. Elliot Hong, L. Elliot Hong, M.D., University of Maryland, Baltimore
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: HP-00044959; 1P50MH082999-01 (NIH)
Record Dates: First submitted 2010-01-04; First posted 2010-04-09 (Estimated); Results first posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-05

CONDITIONS: Schizophrenia
Keywords: Galantamine; Schizophrenia; working memory; cognitive
MeSH Terms: conditions — Schizophrenia | interventions — Galantamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Galantamine, then Placebo (Experimental): Participants took lead-in 3 days of 4mg/ twice a day of galantamine followed by 8 mg on the 4th day, the day of testing. Then, after a period of at least one month, participants took lead-in 3 days of 4mg/ twice a day of placebo followed by 8 mg on the 4th day, the day of testing.
  Interventions: Drug: Galantamine; Drug: Placebo
- Placebo, then Galantamine (Experimental): Participants took lead-in 3 days of 4mg/ twice a day of placebo followed by 8 mg on the 4th day, the day of testing. Then, after a period of at least one month, participants took lead-in 3 days of 4mg/ twice a day of galantamine followed by 8 mg on the 4th day, the day of testing.
  Interventions: Drug: Galantamine; Drug: Placebo

INTERVENTIONS:
Drug: Galantamine — A lead-in 3 days of 4mg/ twice a day of galantamine (or placebo) followed by 8 mg (or placebo) on the 4th day, the day of testing.
  Other Names: Razadyne; 01RZ437
Drug: Placebo — Subjects will be randomly assigned to the two possible order of administration: the drug and then placebo, or the placebo and then drug. Subjects will be given a lead-in 3 days of 4mg/ twice a day of galantamine (or placebo) followed by 8 mg (or placebo) on the 4th day, the day of testing.

SUMMARY:
Schizophrenia is a chronic disorder with onset of psychosis occurring in late teen early twenties, with cognitive impairments and negative symptoms frequently emerging much earlier. Such cognitive impairments and negative symptoms but much milder are also observed in high-risk groups (such as relatives of schizophrenia patients), who may or may not develop the full blown psychotic disorder. Our study plans to recruit such non-ill subjects to test the effects of galantamine on clinical/physiological/cognitive measures. This study serves several goals: If a drug is found effective in treating subtle deficits, then it will provide treatment strategy in individuals with schizophrenia spectrum personality disorders and for early intervention in schizophrenia. In addition, one of the difficulties of testing a drug on schizophrenia is that patients take other medications (i.e., antipsychotic drugs) that can change the effects of the test drug. The proposed study will be in subjects who will not be taking antipsychotic medications. Our study will be carried out in two sessions, at least one month apart. Subjects will be randomly assigned to the two possible order of administration: the drug and then placebo, or the placebo and then drug. Subjects will be given a lead-in 3 days of 4mg/ twice a day of galantamine (or placebo) followed by 8 mg (or placebo) on the 4th day, the day of testing. We will administer a battery of clinical/cognitive/neurophysiological tests after the 8 mg drug dose.

ELIGIBILITY:
Inclusion Criteria:

* age range of 18-64 (confirmed by drivers license or other form of identification)
* the presence of 3 or more SSP symptoms (at least 2 of the SSP symptoms will be negative symptoms as defined by the schizoid traits)
* the presence of visuospatial working memory impairment as defined by error in the oculomotor delayed response (ODR) task of more than 0.5 SD above the mean values in healthy control subjects
* relative of an individual with schizophrenia, schizoaffective disorder, or schizophreniform disorder
* able to provide written informed consent (ESC score 10 or above)

Exclusion Criteria:

* subjects meeting criteria for a life-time diagnosis of any one of the DSM IV, Axis I psychotic disorders (exceptions being a single past episode of major depressive disorder with psychotic features or psychotic symptoms associated with substance abuse with the substance abuse ending 6-months prior to study participation) (this is for the SSP recruitment)
* subjects meeting DSM-IV criteria for current alcohol or substance dependence (other than nicotine) within the last 6 months or DSM-IV criteria for alcohol or substance abuse (other than nicotine) within the last month
* medical conditions that preclude participation in drug trials or assessments of outcome measures (including significant brain, cardiac, liver, lung, endocrinological or metabolic disorders)
* received any investigational drug in the preceding four weeks
* pregnant or of childbearing age and not using a medically approved form of birth control

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2010-05; Primary Completion 2014-08-21 (Actual); Study Completion 2014-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: L. E. Hong, M.D., Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland, Baltimore, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Galantamine, Then Placebo | Placebo, Then Galantamine
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All participants that were included in the study
Arm/Group | All Study Participants
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.33 (5.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 2
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: RVIP Target Hit and False Alarm (Number of Responses)
Description: Rapid Visual Information Processing (RVIP) measures primarily sustained attention but perhaps also working memory. The task was continuous stimuli presentation of a stream of single digits (from 1 to 9) presented in the center of the computer monitor at a rate of 1/600milliseconds; the subjects respond when the they see a target sequence of 3 odds or 3 evens in consecutive sequence. Two target sequences are separated by a minimum and maximum of 30 non-target digits.
Time Frame: 25 minutes (duration needed to complete this test)
Population: Analyzable data for all participants was not available
Measure: Mean (Standard Deviation); unit: Number of responses
Groups:
- Galantamine: Participants took lead-in 3 days of 4mg/ twice a day of galantamine followed by 8 mg on the 4th day, the day of testing.
- Placebo: Participants took lead-in 3 days of 4mg/ twice a day of placebo followed by 8 mg on the 4th day, the day of testing.
Arm/Group | Galantamine | Placebo
Number analyzed (Participants) | 10 | 9
Number of responses
  RVIP Practice Mean Target Hits | 23.4 (6.5) | 22.8 (7.47)
  RVIP Practice Mean False Alarms | 19.7 (18.91) | 14.88 (18.12)
  RVIP First Half Mean Target Hits | 25.4 (8.11) | 19.75 (5.42)
  RVIP First Half Mean False Alarms | 20.7 (19.24) | 18.88 (26.49)
Statistical Analysis 1: Comparison: Galantamine vs Placebo; Comparison of RVIP Practice Mean Target Hits between Galantamine and Placebo Arms; Test type: Superiority; p = 0.898, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Galantamine vs Placebo; Comparison of RVIP Practice Mean False Alarms between Galantamine and Placebo Arms; Test type: Superiority; p = 0.701, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Galantamine vs Placebo; Comparison of RVIP First Half Mean Target Hits between Galantamine and Placebo Arms; Test type: Superiority; p = 0.16, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Galantamine vs Placebo; Comparison of RVIP First Half Mean False Alarms between Galantamine and Placebo Arms; Test type: Superiority; p = 0.701, Wilcoxon (Mann-Whitney)

2. Primary Outcome: RVIP Reaction Times (ms)
Description: as for outcome 1
Time Frame: 25 minutes (total duration to test RVIP)
Population: Analyzable data for all participants was not available
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Galantamine | Placebo
Number analyzed (Participants) | 10 | 9
milliseconds
  RVIP Practice Mean Target Reaction Time | 534.2 (63.3) | 581.5 (82.1)
  RVIP Practice Mean False Alarm Reaction Time | 290.5 (67.5) | 380.5 (75.4)
  RVIP First Half Mean Target Reaction Time | 525.1 (58.7) | 544 (105.6)
  RVIP First Half Mean False Alarm Reaction Time | 215 (129) | 260 (104)
Statistical Analysis 1: Comparison: Galantamine vs Placebo; Comparison of RVIP Practice Mean Target Reaction Time between Galantamine and Placebo Arms; Test type: Superiority; p = 0.161, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Galantamine vs Placebo; Comparison of RVIP Practice Mean False Alarm Reaction Time between Galantamine and Placebo Arms; Test type: Superiority; p = 0.028, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Galantamine vs Placebo; Comparison of RVIP First Half Mean Target Reaction Time between Galantamine and Placebo Arms; Test type: Superiority; p = 0.899, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Galantamine vs Placebo; Comparison of RVIP First Half Mean False Alarms Reaction Time between Galantamine and Placebo Arms; Test type: Superiority; p = 0.521, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Trust Game (Dollar Amount Earned)
Description: Participants compete in a social trust game in which they are paired with a partner (the computer program). Over the course of 24 rounds he participant can offer up to $10 to their partner. The partner can either accept the offer, in which case the total amount offered is split equally between the participant and their partner (i.e. $10 is split into $5 each). Or the partner can reject the offer and receive a portion of the toal offer for themselves and give the participant nothing ($0). The total amount of money that can be offered ranges from $0-240.
Time Frame: 20 minutes (total duration of the trust game cognitive test)
Population: Analyzable data for all participants was not available
Measure: Mean (Standard Deviation); unit: Dollars
Arm/Group | Galantamine | Placebo
Number analyzed (Participants) | 10 | 9
Dollars | 147.7 (81.1) | 131.4 (42.3)
Statistical Analysis 1: Comparison: Galantamine vs Placebo; Comparison of the mean total amount offered during the trust game between the galantamine and placebo groups; Test type: Superiority; p = 0.67, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Brief Assessment of Cognition for Schizophrenia (BACS) Score
Description: The BACS Symbol Coding subtest will be used to assess processing speed, and the demographically corrected T score, will be used for data analysis. This test requires less than 5 minutes to administer adn provides a highly reliable measure of processing speed. There are nine symbols coded 1 through 9. Participants are given 90 seconds to match a series of these symbols with their corresponding number. The total correct matches in the participants score. Scores range from 0-110.
Time Frame: 5 minutes (duration needed to complete the assessment)
Population: Analyzable data for all participants was not available
Measure: Mean (Standard Deviation); unit: Number of correct responses
Arm/Group | Galantamine | Placebo
Number analyzed (Participants) | 10 | 9
Number of correct responses | 49 (9.82) | 52 (8)
Statistical Analysis 1: Comparison: Galantamine vs Placebo; Comparison of the mean correct responses between galantamine and placebo; Test type: Superiority; p = 0.32, Wilcoxon (Mann-Whitney)

5. Primary Outcome: Hopkins Verbal Learning Test (HVLT) Score
Description: HVLT comes in 6 different forms. Forms 4 and 5 were used for this study with one form administered on the first day and the other on the second and were counterbalanced between subjects. Each form contains 12 nouns, four words each from one of three semantic categories, to be learned over the course of three learning trials.
Time Frame: 15 minutes (duration needed to complete this test)
Population: Analyzable data for all participants was not available
Measure: Mean (Standard Deviation); unit: Number of correct responses
Arm/Group | Galantamine | Placebo
Number analyzed (Participants) | 10 | 9
Number of correct responses
  HVLT Trial 1 | 7.7 (2.26) | 7.22 (1.99)
  HVLT Trial 2 | 9.7 (1.77) | 10.22 (1.48)
  HVLT Trial 3 | 10.8 (1.55) | 10.78 (1.3)
Statistical Analysis 1: Comparison: Galantamine vs Placebo; Comparison of the number of correct response on Trial 1 between galantamine and placebo; Test type: Superiority; p = 0.659, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Galantamine vs Placebo; Comparison of the number of correct response on Trial 2 between galantamine and placebo; Test type: Superiority; p = 0.541, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Galantamine vs Placebo; Comparison of the number of correct response on Trial 3 between galantamine and placebo; Test type: Superiority; p = 0.838, Wilcoxon (Mann-Whitney)

6. Primary Outcome: Reading the Mind in the Eyes Score (Number of Correct Responses)
Description: A 30 item task presents a picture of a person's eyes and the participant is asked to determine the person's mental state from 4 multiple choice options.
Time Frame: 10 minutes (duration needed to complete the test)
Population: Analyzable data was not available for all participants
Measure: Mean (Standard Deviation); unit: Number of correct responses
Arm/Group | Galantamine | Placebo
Number analyzed (Participants) | 10 | 9
Number of correct responses | 24.9 (5.26) | 24.12 (3.98)
Statistical Analysis 1: Comparison: Galantamine vs Placebo; A comparison the mean correct responses between galantamine and placebo; Test type: Superiority; p = 0.548, Wilcoxon (Mann-Whitney)

7. Primary Outcome: The Brief Smell Identification Test (B-SIT) Score (Number of Correct Responses)
Description: The Brief Smell Identification Test (B-SIT) is a 5-minute, 12-item screening test. Participants try to identify 12 different odors with four multiple choice options given for each odor.
Time Frame: 5 minutes (duration usually needed to complete this test)
Population: analyzable data for all participant was not available
Measure: Mean (Standard Deviation); unit: Number of correct responses
Arm/Group | Galantamine | Placebo
Number analyzed (Participants) | 10 | 9
Number of correct responses | 10.2 (1.476) | 10.222 (0.833)
Statistical Analysis 1: Comparison: Galantamine vs Placebo; Test type: Superiority; p = 0.871, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Social Affiliation Measured by Social Affiliative Role Play (Rating Scale Score)
Description: In a videotaped session, research staff engages the participant in social interaction based on a role play. The tape is rated on social skills and on Positive and Negative Affect Scale. participants are rated on a 5 point likert scale ranging from very poor (1) to very good (5)
Time Frame: 30 minutes (time needed to complete this test)
Population: analyzable data was not available for all participants
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Galantamine | Placebo
Number analyzed (Participants) | 10 | 10
units on a scale
  Overall Affect | 3.958 (0.68) | 3.8 (0.632)
  Overall Social Skill | 4.15 (0.58) | 3.8 (0.715)
Statistical Analysis 1: Comparison: Galantamine vs Placebo; Comparison of Overall Affect between galantamine and placebo; Test type: Superiority; p = 0.626, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Galantamine vs Placebo; Comparison of Overall Social Skill between galantamine and placebo; Test type: Superiority; p = 0.234, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Facial Affect Recognition Score (Number of Responses)
Description: This computer administered test includes 40 color photogralhs of four emotions (happy, sad, angry, and fearful) balanced for the posers gender, age and ethnicity, including four low intensity and four high intensity facila expressions of each emotion, plus 8 neutral faces. The stimuli are presented in random order and subjects are asked to identify which stimuli were presented to them at the end. Performance on this test correlates with negative symptom severity
Time Frame: 10 minutes (time usually needed to complete this test)
Population: analyzable data was not available for all participants
Measure: Mean (Standard Deviation); unit: Number of Responses
Arm/Group | Galantamine | Placebo
Number analyzed (Participants) | 10 | 9
Number of Responses
  Facial Affect Total | 31.2 (4.49) | 33 (5.21)
  Facial Affect Hits | 12.3 (7.07) | 14.38 (4.75)
  Facial Affect False Alarms | 5.1 (4.46) | 5.38 (3.07)
Statistical Analysis 1: Comparison: Galantamine vs Placebo; Comparison of Facial Affect Total Responses between galantamine and placebo; Test type: Superiority; p = 0.797, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Galantamine vs Placebo; Comparison of Facial Affect Total Hits between galantamine and placebo; Test type: Superiority; p = 0.669, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Galantamine vs Placebo; Comparison of Facial Affect Total False Alarms between galantamine and placebo; Test type: Superiority; p = 0.668, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Collected over the course of 2 approximately 8 hour study days
Description: The Side Effect Checklist was used
Arm/Group | Galantamine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 4/12 | 1/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Galantamine (N=12) | Placebo (N=12)
Dizziness (General disorders) | 2 (2) | 0 (0) — Participant reported felling dizzy after taking study medication or placebo
Euphoria (General disorders) | 1 (1) | 0 — Participant reported felling euphoric during testing
Drowsiness (General disorders) | 1 (1) | 0 (0) — Participant reported feeling drowsy during testing
Blurred Vision (General disorders) | 1 (1) | 0 (0) — Participant reported blurry vision during testing
Tearing of Eyes (General disorders) | 1 (1) | 0 (0) — Participant reported tearing in their eyes during testing
Insomnia (General disorders) | 2 (2) | 0 (0) — Participant reported difficulty sleeping after starting study medication or placebo
Nausea (General disorders) | 2 (2) | 0 (0) — Participant reported felling nauseous after starting study medication or placebo
Headache (General disorders) | 1 (1) | 1 (1) — Participant reported headache after starting study medication or placebo
Malaise (General disorders) | 1 (1) | 0 (0) — Participant reported malaise/physical fatigue after starting study medication or placebo
Sedation (General disorders) | 1 (1) | 0 (0) — Participant reported sedation after starting study medication or placebo
Dry mouth (General disorders) | 1 (1) | 0 (0) — Participant reported dry mouth after starting study medication or placebo
Abdominal Pain (General disorders) | 1 (1) | 0 — Participant reported abdominal pain after starting study medication or placebo

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No